CLINICAL TRIAL: NCT05761301
Title: A Phase 1/2, Randomized, Double-blind, Placebo-controlled, 2-Part Study of the Safety, Tolerability, Efficacy, Pharmacokinetics, and Pharmacodynamics of Single Dose ALN-KHK in Overweight to Obese Adult Healthy Volunteers and Multiple Dose ALN-KHK in Obese Patients With Type 2 Diabetes Mellitus (T2DM)
Brief Title: A Phase 1/2 Study to Evaluate ALN-KHK in Overweight to Obese Healthy Volunteers and Obese Patients With T2DM
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business reasons (not safety related)
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: ALN-KHK-001
Record Dates: First submitted 2023-02-24; First posted 2023-03-09 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Overweight; Obese; Fructose; siRNA; HbA1C; Insulin; Glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: The single ascending dose part of this study (Part A) will have a sequential interventional study model. The multi-dose part of this study (Part B) will have a parallel interventional study model and will begin after the completion of Part A.
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: ALN-KHK (Experimental): Participants will be administered a single dose of ALN-KHK.
  Interventions: Drug: ALN-KHK
- Part A: Placebo (Placebo Comparator): Participants will be administered a single dose of placebo.
  Interventions: Drug: Placebo
- Part B: ALN-KHK (Experimental): Participants will be administered a multiple doses of ALN-KHK.
  Interventions: Drug: ALN-KHK
- Part B: Placebo (Placebo Comparator): Participants will be administered a multiple doses of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALN-KHK — ALN-KHK will be administered by subcutaneous (SC) injection.
  Arms: Part A: ALN-KHK; Part B: ALN-KHK
Drug: Placebo — Placebo will be administered by subcutaneous (SC) injection.
  Arms: Part A: Placebo; Part B: Placebo

SUMMARY:
To evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of single ascending doses of ALN-KHK and to evaluate the safety, tolerability, efficacy, PK and PD of multiple doses of KHK.

ELIGIBILITY:
Inclusion Criteria:

* Stable euthyroid status (no known changes in thyroid function; stable hormone replacement for at least 4 months) at screening
* Part A: body mass index (BMI) ≥27 kg/m^2 and ≤34.9 kg/m^2
* Part B: BMI ≥30 kg/m^2 to ≤39.9 kg/m^2, confirmed diagnosis of T2DM, and an HbA1c ≥7.5% to <10%
* Part B: Confirmed T2DM diagnosis

Exclusion Criteria:

* Parts A and B: has received an investigational agent within the last 30 days
* Part A: History of Type 1 or Type 2 diabetes
* Part B: History of Type 1 diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Part A: Frequency of Adverse Events | Up to 9 Months
Part B: Frequency of Adverse Events | Up to 12 Months

SECONDARY OUTCOMES:
Part A: Area Under the Concentration-time Curve (AUC) of ALN-KHK and Potential Major Metabolite(s) | Up to 2 Days following dosing on Day 1
Part A: Maximum Observed Plasma Concentration (Cmax) of ALN-KHK and Potential Major Metabolite(s) | Up to 2 Days following dosing on Day 1
Part A: Time to Maximum Observed Plasma Concentration (Tmax) of ALN-KHK and Potential Major Metabolite(s) | Up to 2 Days following dosing on Day 1
Part A: Fraction of ALN-KHK Excreted in the Urine (fe) and Potential Major Metabolite(s) | Postdose on Day 1
Part A: Percent Change from Baseline in Circulating Fructose in Response to a Fructose Tolerance Test | Baseline up to Month 6
Part A: Percent Change from Baseline in Urinary Fructose in Response to a Fructose Tolerance Test | Baseline up to Month 6
Part A: Percent Change from Baseline in Circulating Fibroblast Growth Factor 21 (FGF21) in Response to a Fructose Tolerance Test | Baseline up to Month 6
Part B: Absolute Change from Baseline in Hemoglobin A1C (HbA1c) at 6 Months | Baseline and Month 6
Parts A and B: Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) in Response to a Glucose Tolerance Test | Part A: Screening up to Month 3; Part B: Month 4
Part B: Fasting Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) | Month 4
Parts A and B: Glucose and Insulin AUC in response to Tolerance Test | Part A: Screening up to Month 3; Part B: Month 4
Part B: Plasma Concentrations of ALN-KHK and Potential Major Metabolite(s) | Day 1 and Month 3

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (15):
- United States (11):
  - Clinical Trial Site, Phoenix, Arizona
  - Clinical Trial Site, Vista, California
  - Clinical Trial Site, Lake Worth, Florida
  - Clinical Trial Site, Orlando, Florida
  - Clinical Trial Site, Atlanta, Georgia
  - Clinical Trial Site, Berlin, New Jersey
  - Clinical Trial Site, Monroe, North Carolina
  - Clinical Trial Site, Oklahoma City, Oklahoma
  - Clinical Trial Site, Dallas, Texas
  - Clinical Trial Site, Houston, Texas
  - Clinical Trial Site, San Antonio, Texas
- Canada (4):
  - Clinical Trial Site, Sarnia, Ontario
  - Clinical Trial Site, Montreal, Quebec
  - Clinical Trial Site, Victoriaville, Quebec
  - Clinical Trial Site, Toronto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Badri P, Kolachana K, Duong A, Lasko M, Nandi T, Mehrotra N, Robbie GJ. Platform Assessment of Concentration-QTc Relationship Across GalNAc-siRNA Molecules. Clin Pharmacokinet. 2025 Dec 12. doi: 10.1007/s40262-025-01606-0. Online ahead of print. PMID 41388232